CLINICAL TRIAL: NCT01904422
Title: Evaluation of the Effectiveness of Intensive Periodontal Treatment as Compared to Conventional Periodontal Treatment on the Level of Glycosylated Hemoglobin in Patients With Decompensated Type 2 Diabetes Mellitus: Randomized Clinical Trial
Brief Title: Periodontal Treatment in Non-controlled Type 2 Diabetes Mellitus Patients. Clinical Trial
Acronym: FONIS12I2106
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Dr. Antonio Quintero, Professor of Periodontics Department, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Universidad de los Andes
Record Dates: First submitted 2013-07-14; First posted 2013-07-22 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus.; Chronic Periodontitis
Keywords: Diabetes mellitus.; Periodontitis; Periodontal treatment.
MeSH Terms: conditions — Diabetes Mellitus; Chronic Periodontitis; Periodontitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional periodontal treatment (Experimental): Treatment group by quadrant in five weeks. Patients in this group will receive periodontal treatment including plaque control instructions, supragingival and subgingival debridement and root planing. This treatment is done in 5 sessions with a periodicity of 1 session per week. In the first session patients will receive hygiene instruction and supragingival debridement performed with and ultrasonic device. In the following session, there will be done the scaling and root planing to one quadrant per session, using site specific hand curettes. In case of being partially edentulous patients will be implemented at least 3 teeth per quadrant in each session.
  Interventions: Procedure: conventional periodontal treatment
- Intensive periodontal treatment (Experimental): Intensive treatment group in 24 hours: Patients in this group will receive periodontal treatment including: plaque control instructions, supragingival and subgingival debridement and scaling and root planing. This treatment is carried out in 2 sessions within 24 hours. In the first session hygiene instruction and supragingival and scaling and root planing of the teeth in right side at the upper jaw and mandible will be performed. The implementation of each upper and lower hemiarcade will be made until the periodontist treating check manually the removal of all subgingival calculus deposit and feel the smoothness of the root surface. In the second session, there will be an identical procedure in the arch left.
  Interventions: Procedure: conventional periodontal treatment

INTERVENTIONS:
Procedure: conventional periodontal treatment
  Other Names: intensive periodontal treatment

SUMMARY:
Periodontitis is an infectious disease that destroys the tooth supporting tissues and triggers a local and systemic immune response. Type 2 Diabetes Mellitus (DM2) is a risk factor for periodontitis.Patients with DM2 and periodontitis have greater difficulty getting and maintaining an appropriate glycemic control. It has been reported an average decrease of 0.4% in glycosylated hemoglobin levels (HbA1c) in patients periodontally treated versus untreated. It is not has been established that periodontal treatment type in spaced sessions (multiple sessions over a period of 4 weeks) or rapid and intensive (2 sessions in 24 hours), has a greater impact on glycemic control in type 2 diabetes patients.

Objective: To evaluate the effectiveness of intensive periodontal treatment modality as compared with conventional on HbA1c level in periodontitis and DM2 decompensated patients.

DETAILED DESCRIPTION:
It is proposed to conduct a clinical trial in 100 type 2 diabetic patients with poor glycemic control defined as a glycated hemoglobin (HbA1c) ≥ 7% at last check, with randomization stratified by referral center, with two parallel groups (1: 1). Diabetic patients are in treatment and control in Diabetes Polyclinic Medical Specialty Center of the University of the Andes or the medical polyclinic Joan Alsina in San Bernardo . All decompensated DM2 patients diagnosed with chronic periodontitis will receive periodontal treatment based on 2 different periodontal treatment modalities: the first and most traditional is by spaced sessions by quadrant in 1 weekly session (5 sessions). The second form of treatment corresponds to an intensive periodontal treatment, whole mouth in 24 hours.

All patients will be given an initial periodontal examination with manual north carolina periodontal probe, performed by a single operator previously calibrated.

Periodontal status will be determine according to the classification of Page and Eke (2007) and periodontal wound size (PISA) will be also determine. Also, will be measured inflammatory mediators and cytokines in both plasma and gingival crevicular fluid (GCF) by ELISA test. The data were entered into a medical record designed specifically for this study and the variables will be recorded prior and at 3 and 6 months after periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated type 2 diabetic patients (HbA1c ≥ 7% at last check).
* Minimum 12 teeth in the mouth.
* no history of surgical or nonsurgical periodontal treatment in the six months prior to baseline.
* not be involved in another clinical trial.

Exclusion Criteria:

* Patients with renal failure
* Patients with rheumatoid arthritis,
* Patients with heart disease.
* Patients with history of stroke or acute cardiovascular event in the 12 months prior to the start of the study.
* Patients with liver dysfunction
* Patients in state of pregnancy or planning pregnancy.
* Patients on medical treatment with systemic antibiotics in the past 3 months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | 2 years
  Assess levels and relationship of HbA1c in peripheral blood and gingival crevicular fluid at baseline, 3 and 6 months after periodontal treatment in the group of patients treated by intensive and conventional periodontal treatment.

SECONDARY OUTCOMES:
C-reactive protein | 2 years
  Assess levels and relationship of C-reactive protein, in peripheral blood and gingival crevicular fluid at baseline, 3 and 6 months after periodontal treatment in the group of patients treated by intensive and conventional periodontal treatment .
Interleukin-6 (IL-6) | 2 years
  Assess levels and relationship of IL-6 in peripheral blood and gingival crevicular fluid at baseline, 3 and 6 months after periodontal treatment in the group of patients treated by intensive and conventional treatment.
Tumor Necrosis Factor (TNF) | 2 years
  Asses levels and relationship of TNF in peripheral blood and gingival crevicular fluid at baseline, 3 and 6 months after intensive and conventional periodontal treatment.

OTHER OUTCOMES:
probing depth | 2 years
  Asses the levels of probing depth baseline, 3 and 6 months after periodontal treatment in the group of patients treated by intensive and conventional treatment.
gingival bleeding (BOP) | 2 years
  Asses the level of BOP at baseline, 3 and 6 months after periodontal treatment in both groups of patients.
clinical attachment level (CAL) | 2 years
  Asses the level of CAL baseline, 3 and 6 months after periodontal treatment in the group of patients treated by intensive and conventional treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J Quintero, DDS, Principal Investigator — Universidad de Los Andes
Locations (1):
- Joan Alsina Polyclinic, San Bernardo, Metropolitan, Chile

REFERENCES:
- [Derived] Quintero AJ, Chaparro A, Quirynen M, Ramirez V, Prieto D, Morales H, Prada P, Hernandez M, Sanz A. Effect of two periodontal treatment modalities in patients with uncontrolled type 2 diabetes mellitus: A randomized clinical trial. J Clin Periodontol. 2018 Sep;45(9):1098-1106. doi: 10.1111/jcpe.12991. Epub 2018 Aug 16. PMID 30024030